CLINICAL TRIAL: NCT00846001
Title: Study of Resynchronization and CABG Unified Efficacy in Ischemic Heart Failure Patients
Brief Title: Resynchronization Surgery Combined Unified Efficacy
Acronym: RESCUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Collaborators: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SACRT 022; RU 001
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Ischemic Heart Failure
Keywords: Resynchronization Therapy
MeSH Terms: interventions — Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CABG alone (Active Comparator): Standard coronary artery bypass grafting according guidelines
  Interventions: Procedure: Coronary artery bypass grafting
- CABG+CRT (Experimental): Standard coronary artery bypass grafting according guidelines with concomitant three bipolar epicardial leads implantation for cardiac resynchronization therapy
  Interventions: Procedure: Coronary artery bypass grafting; Device: Epicardial implantation of cardiac resynchronization therapy device

INTERVENTIONS:
Procedure: Coronary artery bypass grafting — Standard coronary surgry according guidelines
Device: Epicardial implantation of cardiac resynchronization therapy device — During the cardiac surgery, the CABG+CRT arm patients will be implanted with epicardial leads to the right atrium, right and left ventricles. Left ventricle leads will be fixed to the posterolateral wall provided that there is no scar or fat tissue (behind and 2-3 cm apical than obtuse marginal artery). Right atrial and right ventricular leads will be fixed in a traditional way. Then the leads will be guided into a preformed pocket (left subclavian region) and connected with the CRT device.
  Arms: CABG+CRT

SUMMARY:
The purpose of the study is to compare survivability and efficacy of the patients with severe ischemic heart failure after coronary artery bypass grafting alone and coronary artery bypass grafting with single-step implantation of CRT system (CABG alone vs CABG + CRT )

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Age 18-80
* History of ischemic heart failure and indications for CABG
* LVEF less than 35% estimated by echocardiography measured within 3 months of study entry
* NYHA and CCS (angina) II-IV functional class
* Signs of dyssynchrony (at least one of the following three): QRS > 120 ms or dyssynchrony based on Doppler-methods (Tissue Tracking and TSI methods) or CARE HF criteria: Aortic pre-ejection delay >140ms, Interventricular mechanical delay >40 ms, Delayed activation of postero-lateral LV wall

Exclusion Criteria:

* Failure to provide informed consent.
* Previous cardiac surgery
* Non-cardiac illness with a life expectancy of less than 3 year
* Non-cardiac illness imposing substantial operative mortality
* Previous heart, kidney, liver, or lung transplantation
* Current participation in another clinical trial in which a patient is taking an investigational drug or receiving an investigational medical device
* Successful coronary revascularization (СABG or PCI) within 12 months of study enrollment
* Chronic atrial fibrillation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Long-term mortality | 6 years

SECONDARY OUTCOMES:
Mode of Death | 6 years
Adverse cardiac events | 6 years
Lead performance | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny A Pokushalov, MD, PhD, Prof., Principal Investigator — State Research Institute of Circulation Pathology
Locations (3):
- Medical University of Silesia, Katowice, Poland
- State Research Institute of Circulation Pathology, Novosibirsk, Russia
- University Medical Center, Ljubljana, Slovenia

REFERENCES:
- [Result] Pokushalov E, Romanov A, Prohorova D, Cherniavsky A, Goscinska-Bis K, Bis J, Bochenek A, Karaskov A. Coronary artery bypass grafting with concomitant cardiac resynchronisation therapy in patients with ischaemic heart failure and left ventricular dyssynchrony. Eur J Cardiothorac Surg. 2010 Dec;38(6):773-80. doi: 10.1016/j.ejcts.2010.03.036. Epub 2010 May 6. PMID 20447832
- [Result] Pokushalov E, Romanov A, Prohorova D, Cherniavsky A, Karaskov A, Gersak B. Coronary artery bypass grafting with and without concomitant epicardial cardiac resynchronization therapy in patients with ischemic cardiomyopathy: a randomized study. Heart Surg Forum. 2010 Jun;13(3):E177-84. doi: 10.1532/HSF98.20091149. PMID 20534420
- [Derived] Romanov A, Goscinska-Bis K, Bis J, Chernyavskiy A, Prokhorova D, Syrtseva Y, Shabanov V, Alsov S, Karaskov A, Deja M, Krejca M, Pokushalov E. Cardiac resynchronization therapy combined with coronary artery bypass grafting in ischaemic heart failure patients: long-term results of the RESCUE study. Eur J Cardiothorac Surg. 2016 Jul;50(1):36-41. doi: 10.1093/ejcts/ezv448. Epub 2015 Dec 30. PMID 26719401